CLINICAL TRIAL: NCT03723915
Title: A Phase 2 Study of Pembrolizumab in Combination With Pelareorep in Patients With Advanced Pancreatic Adenocarcinoma
Brief Title: Pembrolizumab and Pelareorep in Treating Patients With Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The total accrual goal of 34 patients was not met. Stage 1 of the study did not meet the interim analysis criteria to move onto Stage 2 of the Simon 2 stage design.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 18I01; NCI-2018-02319 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00207577; NU 18I01 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, wild-type reovirus) (Experimental): See Detailed Description
  Interventions: Biological: Pembrolizumab; Biological: Wild-type Reovirus

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Wild-type Reovirus — Given pelareorep IV
  Other Names: Reolysin

SUMMARY:
This phase II trial studies the side effects and how well pembrolizumab in combination with pelareorep work in treating patients with pancreatic cancer that has spread to other parts of the body. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. A virus, called reovirus (pelareorep), which has been changed in a certain way, may be able to kill tumor cells without damaging normal cells. Giving pembrolizumab in combination with pelareorep may work better in treating patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria of pembrolizumab in combination with Reovirus Serotype 3 ? Dearing Strain (pelareorep).

SECONDARY OBJECTIVES:

I. To determine progression free survival by RECIST v 1.1 criteria, as well as 1- year, 2-year and median overall survival with pembrolizumab in combination with pelareorep.

II. To determine safety and tolerability of pembrolizumab and pelareorep when administered in combination as determined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.03.

III. To determine the effects (immune response) of pembrolizumab and pelareorep when administered in combination as determined by analysis of pre-and post-treatment biopsies and blood-based immune markers.

EXPLORATORY OBJECTIVES:

I. To measure the overall response rate (ORR) by using Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST) criteria, for the combination of pembrolizumab and pelareorep.

II. To determine progression free survival by iRECIST criteria as well as 1-year, 2-year and median overall survival with pembrolizumab in combination with pelareorep.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 32 courses in the absence of disease progression, unacceptable toxicity, development of an inter-current illness that prevents further administration of treatment, patient decides to withdraw, patients not experiencing clinical benefit in the judgment of the Investigator, or the treating investigator determines that the patient should be taken off treatment for any reason. Patients also receive Pelareorep IV over 60 minutes on days 1, 2, 3, and 8 in course 1 and on days 1 and 8 of subsequent courses. Courses repeat every 21 days for up to 24 months in the absence of disease progression, unacceptable toxicity, development of an inter-current illness that prevents further administration of treatment, patient decides to withdraw, patients not experiencing clinical benefit in the judgment of the Investigator, or the treating investigator determines that the patient should be taken off treatment for any reason. Patients who stop study therapy with stable disease (SD) or better may be eligible for up to 1 year of additional Pelareorep and pembrolizumab therapy if they progress after stopping study treatment.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced (unresectable or metastatic) pancreatic adenocarcinoma, documented objective radiographic progression and have failed or not tolerated first-line therapy.

  * Note: First-line therapy denotes systemic chemotherapy for advanced pancreatic adenocarcinoma. Only one line of therapy is permitted in this setting. Intolerant to first line therapy are patients that have developed >= grade 3 adverse events related to first line therapy and treating physician deems continuing of systemic chemotherapy would be detrimental to patient.
* Patients must have confirmation of an existing formalin-fixed paraffin-embedded (FPPE) tumor sample from archival tissue or from a fresh biopsy of a primary or metastatic lesion at baseline, either as a block or unstained slides for performance of correlative studies.

  * Note: Patients must undergo a fresh biopsy if archival tissue is not available.
* Patients must have measurable disease as defined by RECIST v 1.1.
* Any major surgery (except biopsies) must have occurred at least 28 days prior to first day of study treatment.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance score =< 1.
* Patients must have a life expectancy of >= 6 months.
* Absolute neutrophil count (ANC) >= 1,500 /mcL (with or without growth factor use).
* Platelets >= 100,000 / mcL.
* Hemoglobin >= 9 g/dL, OR >= 5.6 mmol/L with (if clinically indicated)/without transfusion or erythropoietin [EPO] dependency).
* Serum creatinine =< 1.5 x upper limit of normal (ULN), OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN.

  * (Note: creatinine clearance should be calculated per institutional standard.)
* Serum total bilirubin =< 1.5 x ULN, OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN, OR =< 5 x ULN for subjects with liver metastases.
* Albumin >= 2.5 mg/dL.
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy. For patients on anticoagulant therapy, PT/INR must be within therapeutic range.
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy. For patients on anticoagulant therapy, PT/INR must be within therapeutic range
* Thyroid-stimulating hormone (TSH), thyroxine (T4) and corticotropin (ACTH) within normal range (prior to registration).
* Proteinuria within institutional normal or =< grade 1 OR urinary protein < 1 g/24 hours (hr) (prior to registration).
* Female subject of childbearing potential must have a negative urine or serum pregnancy within 7 days of registration. It is to be repeated on day 1 of study treatment, before infusion, if it is done greater than 3 days of day 1. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required. Female subjects of childbearing potential must be willing to use an adequate method of contraception (willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity), for the course of the study through 120 days after the last dose of study medication. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  * Note: A female of childbearing potential (FOCBP) is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months).
* Male subjects of childbearing potential must agree to use an adequate method of contraception or be surgically sterile or abstain from heterosexual activity, starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Patients must have signed an informed consent indicating that the patient is aware of the neoplastic nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
* Patients must be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior first day of study drug or those who have not recovered from adverse events due to agents administered more than 4 weeks from cycle 1 day 1 are not eligible.
* Patients who have a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment are excluded.

  * Note: If patient is on high dose of steroid therapy, it needs to be brought down to < 10 mg prednisone or equivalent for at least 7 days prior to day 1 of study treatment.
* Patients receiving any other investigational agents for at least 4 weeks before the first dose of study treatment are not eligible.
* Patients with a known history of active TB (Bacillus tuberculosis) are excluded.
* Patients with a hypersensitivity to pembrolizumab or any of its excipients are excluded.
* Patients who have had a prior anti-cancer monoclonal antibody (mAb) within 28 days prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Patients who have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 28 days prior to study day 1 or who has not recovered (i.e., NCI CTCAE version 4.03 grade =< 1 or at baseline) from adverse events due to a previously administered agent are not eligible.

  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
  * Exceptions to this criteria are:

    * Subjects with =< grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study.
* Patients receiving palliative radiation are eligible for this study. Palliative radiation is allowed during treatment as well. Patients with a known additional malignancy that is progressing or requires active treatment within the past 5 years are excluded. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Patients with a known active central nervous system (CNS) metastases and/or carcinomatous meningitis are excluded.

  * Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
  * This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Patients with an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs) are excluded.

  * Note: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Patients with a history of (non-infectious) pneumonitis that required steroids or current pneumonitis are excluded.
* Patients with an active infection requiring systemic therapy are excluded.
* Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator are excluded.
* Patients with a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial are excluded.
* Patients who are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment are excluded.
* Patients who have received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PDL2 agent are excluded.
* Patients with a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) are excluded.
* Patients with a known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected) are excluded.
* Patients who have received a live vaccine within 30 days of planned start of study therapy are excluded.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
* Patients with clinically significant cardiac disease (New York Heart Association, class III or IV including pre-existing arrhythmia, uncontrolled angina pectoris, and myocardial infarction 1 year prior to registration, or grade 2 or higher compromised left ventricular ejection fraction are excluded.
* Patients who have dementia or altered mental status that would prohibit informed consent are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2021-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Mahalingam D, Chen S, Xie P, Loghmani H, Heineman T, Kalyan A, Kircher S, Helenowski IB, Mi X, Maurer V, Coffey M, Mulcahy M, Benson A, Zhang B. Combination of pembrolizumab and pelareorep promotes anti-tumour immunity in advanced pancreatic adenocarcinoma (PDAC). Br J Cancer. 2023 Sep;129(5):782-790. doi: 10.1038/s41416-023-02344-5. Epub 2023 Jul 13. PMID 37443348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened up to patient accrual on Nov. 2, 2018 with the first patient starting treatment Nov. 14, 2018 and an accrual goal of 34 patients. Stage 1 of the Simon 2 Stage design was completed on Jan 23, 2020, and the study was closed to accrual. The study did not meet the interim analysis criteria to continue to stage 2. Pharmacodynamic analysis is ongoing to identify biomarkers to predict response from therapy.
Groups:
- Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50: Pembrolizumab will be administered on Day 1 of each cycle at 200 mg IV over 30 minutes.
  In Cycle 1, Pelareorep will be administered at a dose of 4.5x10 ^10 TCID_50 (Tissue Culture Infective Dose 50) over 60 minutes on Days 1, 2, 3 and 8. From Cycle 2 onwards, Pelareorep will be administered at a dose of 4.5x10^10 TCID_50 on Days 1 and 8.
  Pelareorep will be administered after completion of Pembrolizumab infusion on Day 1 of each cycle.
  Each cycle is 21 days (3 weeks). Up to 32 cycles of pembrolizumab and 24 months of Pelareorep (2 years) can be administered in the absence of progression, intolerable toxicity, and other discontinuation criteria (See protocol section 4.6).
Period: Screening
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Started | 17
Completed | 15
Not Completed | 2
Not completed — Failed to meet screening requirements. | 2
Period: On Treatment
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Started | 15
Registered on Study | 15
Received First Dose of Study Drugs | 13
Completed | 13
Not Completed | 2
Not completed — Failed to meet treatment requirements | 2
Period: Survival Follow-up
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Started (Followed until progression (PD) or withdrawal of consent. At PD followed for survival until death.) | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only patients who were treated on study were included. 2 patients were screen fails, and 2 patients became ineligible for treatment and did not receive study drug--these patients were not included here.
Groups:
- Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50: Pembrolizumab will be administered on Day 1 of each cycle at 200 mg IV over 30 minutes.
  In Cycle 1, Pelareorep will be administered at a dose of 4.5x10 ^10 TCID_50 over 60 minutes on Days 1, 2, 3 and 8. From Cycle 2 onwards, Pelareorep will be administered at a dose of 4.5x10^10 TCID_50 on Days 1 and 8.
  Pelareorep will be administered after completion of Pembrolizumab infusion on Day 1 of each cycle.
  Each cycle is 21 days (3 weeks). Up to 32 cycles of pembrolizumab and 24 months of Pelareorep (2 years) can be administered in the absence of progression, intolerable toxicity, and other discontinuation criteria (See protocol section 4.6).
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1
Description: To determine the overall response rate (ORR) by RECIST v 1.1 criteria for the combination of pembrolizumab with pelareorep. ORR is defined as the number of patients who have a complete or partial response to therapy (CR or PR). The Simon 2 stage design for this study requires 2 or more PR or CR in Stage 1 to continue accrual for Stage 2. Per RECIST v. 1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Patients who have taken one dose of either study drug, and completed the first on study scan (last week of Cycle 3) are evaluable. If a patient drops out of the study before the first scan, due to clinical progression, they are evaluable and will not be replaced.
Time Frame: Last week of Cycle 3 (1 Cycle = 21 days)
Population: Although 13 patients received treatment, 1 patient refused treatment after Cycle 1. Their response data was not available for evaluation.
Measure: Number; unit: participants
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Number analyzed (Participants) | 12
participants
  Complete response | 0
  Partial response | 1

2. Secondary Outcome: Median Progression Free Survival (mPFS) by RECIST v 1.1
Description: Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (including baseline if that is the smallest). In addition, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions is also considered progression. Kaplan-Meier curves will be used.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Number analyzed (Participants) | 13
months | 1.8727 [1.6099 to 7.1964]

3. Secondary Outcome: Overall Survival at One Year (12 Months)
Description: Measured from time of treatment initiation until death for any reason. Kaplan-Meier curves will be used.
Time Frame: At 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Number analyzed (Participants) | 13
percentage of patients | 7.69 [1.17 to 50.57]

4. Secondary Outcome: Overall Survival (OS) at Two Years (24 Months)
Description: Measured from time of treatment initiation until death for any reason. Kaplan-Meier curves will be used.
Time Frame: At 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Number analyzed (Participants) | 13
percentage of patients | 7.69 [1.17 to 50.57]

5. Secondary Outcome: Median Overall Survival (OS)
Description: Measured from time of treatment initiation until death from any cause. Kaplan-Meier curves will be used.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Number analyzed (Participants) | 13
months | 6.2094 [2.6270 to 26.0849]

6. Secondary Outcome: Number of Patients With Adverse Events at Grade 3 Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: Adverse events graded 3 using CTCAE 4.03 where:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities.
  Moderate (grade 2): the event causes discomfort that affects normal daily activities.
  Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status.
  Life-threatening (grade 4): the patient was at risk of death at the time of the event.
  Fatal (grade 5): the event caused death.
Time Frame: Up to 30 days after last dose
Measure: Number; unit: patients
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
Number analyzed (Participants) | 13
patients
  Fever | 1
  Vomiting | 1
  Nausea | 1
  Fatigue | 2
  Anemia | 1
  White blood cell decreased | 1
  Alkaline phosphatase increased | 1
  Lymphocyte count decreased | 2
  Neutrophil count decreased | 1
  Hyponatremia | 2

7. Secondary Outcome: Immune Response Determined by Analysis of pre-and Post- Treatment Biopsies and Blood-based Immune Markers
Description: Will be assessed for change using paired statistical methods such as paired t-tests or signed rank tests.
Time Frame: Up to 2 years
Reporting Status: Not Posted, anticipated posting 2023-05

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 2 year period. Each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 30 days post last treatment, where 1 Cycle = 21 days the range of cycles attempted was 1-9.
Description: SAEs are collected from time of consent, and through 30 days post last dose of treatment (thus may include screen-fail patients who did not initiate treatment). All-Cause Mortality and Other Adverse Events are not monitored/assessed for screen-fail patients. Data collection for all-cause mortality and other adverse events begins at the time of treatment initiation.
Arm/Group | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50
All-Cause Mortality (participants affected / at risk) | 11/13
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50 (N=17)
Abdominal Pain (Gastrointestinal disorders) | 2 — * One patient did not receive any study drug--they were included as SAEs are monitored at time of consent. This patient also experienced dehydration at the time of the SAE. * One patient also experienced back pain at the time of this SAE.
Obstruction Gastric (Gastrointestinal disorders) | 3 — One patient also experienced anemia, lymphocyte count decrease, hypoalbuminemia, and nausea at the time of this SAE. One patient also experienced nausea, vomiting, abdominal pain, and duodenal ulcer at the time of this SAE.
Blood bilirubin Increased (Investigations) | 1
Vascular access Complication (RUE DVT) (Injury, poisoning and procedural complications) | 1 — This patient also experienced anemia, bloody stool, and duodenal hemorrhage at the time of this SAE.
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — This patient also experienced stroke at the time of this SAE.
Cholecystitis (Hepatobiliary disorders) | 1 — This patient also experienced fatigue, hyponatremia, nausea, and vomiting at the time of this SAE.
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 — One patient also experienced Death NOS at the time of this SAE.
Endocarditis infective (Infections and infestations) | 1 — This patient also experienced stroke at the time of this SAE.
Constipation (Gastrointestinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 — This patient also experienced depressed level of consciousness, and hypoxia at the time of this SAE. This patient did not receive any study drug. They were included because SAEs are monitored at the time of consent.
Lymphocyte decreased (Investigations) | 1 — This patient also epxerienced nausea, anemia, and hypoalbuminemia at the time of this SAE.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab 200 mg IV + Pelareorep 4.5x10^10 TCID_50 (N=13)
Anemia (Blood and lymphatic system disorders) | 9
Leukocytosis (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 6
Hypothyroidism (Endocrine disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Duodenal stenosis (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastric perforation (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Obstruction gastric (Gastrointestinal disorders) | 3
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Chills (General disorders) | 12
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 10
Fever (General disorders) | 12
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Endocarditis infective (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 5
Cardiac troponin I increased (Investigations) | 1
Fibrinogen decreased (Investigations) | 1
GGT increased (Investigations) | 7
INR increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 8
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 6
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 7
Presyncope (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urine discoloration (Renal and urinary disorders) | 5
Vaginal dryness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 13
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
The total accrual goal of 34 patients was not met. Stage 1 of the study did not meet the interim analysis criteria to move onto Stage 2 of the Simon 2 stage design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03723915/Prot_SAP_000.pdf